CLINICAL TRIAL: NCT00459355
Title: Clinical Trial of a Home Safety Intervention for Alzheimer's Disease
Brief Title: Home Safety Clinical Trial for Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Boston Medical Center (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NRH 05-056
Record Dates: First submitted 2007-04-06; First posted 2007-04-11 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-08

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: Alzheimer's disease; Dementia; Safety; Home Care Services
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home Safety Toolkit (Experimental): Intervention group receives home safety tool-kit with education and self-efficacy materials to promote competence to make home safety modifications.
  Interventions: Behavioral: Home Safety Toolkit
- Conventional Safety Checklist (No Intervention): Comparison group received a conventional home safety checklist

INTERVENTIONS:
Behavioral: Home Safety Toolkit — Health literacy-verified booklet and home safety items to promote competence to make home safety modifications.
  Arms: Home Safety Toolkit

SUMMARY:
The purpose of this study was to test the effectiveness of a new multimodal educational intervention to improve home safety for persons with dementia of the Alzheimer's type and their home caregivers.

DETAILED DESCRIPTION:
Objectives: The purpose of this research study was to test the effectiveness of a new multimodal educational intervention to improve caregiver competence to create a safer home environment, and decrease risk and accidents to veterans with dementia living in the community.

Objective 1: To determine the effect of the Home Safety Toolkit intervention on caregiver self-efficacy, caregiver adherence to home safety recommendations, and caregiver strain.

Objective 2: To determine the effect of the Home Safety Toolkit intervention on the frequency of risky behaviors and accidents among care recipients with dementia of the Alzheimer's type living in the community.

Research Design: This study was a single-blinded clinical trial with random assignment of subjects to either the intervention group that receives the Home Safety Toolkit Intervention or the control group which receives customary care.

Methodology: The sample consisted of primary family caregivers of a person with dementia of the Alzheimer's type (DAT) receiving care at the Bedford VAMC Dementia Outpatient Clinic, the VA Boston HCS, and the Boston University Alzheimer's Disease Center. Subjects were dyads of primary caregivers and persons with a progressive DAT who live in the community, are willing to have home visits for home safety education, and who read and speak English. Inclusion criteria for care recipients were: diagnosis of DAT, score of 24 or less on the Mini-Mental State Exam (MMSE), is expected to continue living in the community for the next 6 months, and has the ability to ambulate without help from the caregiver. Inclusion criteria for the primary informal caregiver were: lives in the home with the care-recipient, provides a minimum of 4 hours of care-giving or supervision per day, and has no known cognitive impairment as judged by the primary care provider who refers the subject dyad for study recruitment. Exclusion criteria were: care-recipient MMSE score of 25 or greater; a previous home safety visit; and admission to a long-term care facility. Persons with DAT who are living alone will be excluded because their safety issues are more complex and there is no primary informal caregiver who can make consistent observations about risky behaviors and accidents. Time 1 and Time 2 data collection was conducted at home visits and interim data collection was done biweekly by phone. A total of 108 subject dyads completed the study, randomly assigned to the control group (N-48 dyads) and intervention group (60 dydads). The length of participation for each caregiver-care recipient dyad was 3 months after which the control group was offered the Home Safety Toolkit. Data analysis used Multivariate Analysis of Covariance (MANCOVA) to test hypotheses for significant group differences with the following outcome variables: adherence to recommendations; post-intervention caregiver self-efficacy and post-intervention caregiver strain; care-recipient risky behaviors and accidents. Covariates will include: baseline measures of caregiver self-efficacy and caregiver strain, caregiver years of formal education and use of social support resources.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are dyads of primary caregivers and persons with a progressive DAT who live in the community, are willing to have home visits for home safety education, and who read and speak English.
* Inclusion criteria for care recipients are: diagnosis of DAT, score of 24 or less on the Mini-Mental State Exam (MMSE), is expected to continue living in the community for the next 6 months, and has the ability to ambulate without help from the caregiver.
* Inclusion criteria for the primary informal caregiver are: lives in the home with the care-recipient, provides a minimum of 4 hours of care-giving or supervision per day, and has no known cognitive impairment as judged by the primary care provider who refers the subject dyad for study recruitment.

Exclusion Criteria:

* Care-recipient MMSE score of 25 or greater.
* A previous home safety visit.
* Admission to a long-term care facility. - Persons with DAT who are living alone will be excluded because their safety issues are more complex and there is no primary informal caregiver who can make consistent observations about risky behaviors and accidents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2007-07; Primary Completion 2010-05 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy J Horvath, PhD RN, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA
Locations (1):
- Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts, United States

REFERENCES:
- [Result] Horvath KJ, Trudeau SA, Rudolph JL, Trudeau PA, Duffy ME, Berlowitz D. Clinical trial of a home safety toolkit for Alzheimer's disease. Int J Alzheimers Dis. 2013;2013:913606. doi: 10.1155/2013/913606. Epub 2013 Sep 29. PMID 24195007
- [Result] Lambe S, Cantwell N, Islam F, Horvath K, Jefferson AL. Perceptions, knowledge, incentives, and barriers of brain donation among African American elders enrolled in an Alzheimer's research program. Gerontologist. 2011 Feb;51(1):28-38. doi: 10.1093/geront/gnq063. Epub 2010 Aug 2. PMID 20679141

RESULTS

PARTICIPANT FLOW:
Groups:
- Checklist: Group receives conventional home safety checklist
Period: Overall Study
Arm/Group | Home Safety Toolkit | Checklist
Started | 140 (Includes 70 dyads, caregiver/care-recipient) | 114 (Includes 57 dyads, caregiver + care-recipient)
Completed | 120 (Includes 60 dyads, caregiver + care-recipient) | 96 (Includes 48 dyads, caregiver + care-recipient)
Not Completed | 20 | 18
Not completed — Subject no longer met inc criteria | 20 | 18

BASELINE CHARACTERISTICS:
Population: Sample size calculations indicated that 216 total participants was sufficient for all calculations
Groups:
- Checklist: Received conventional home safety checklist
- Total: Total of all reporting groups
Arm/Group | Home Safety Toolkit | Checklist | Total
Number analyzed (Participants) | 120 | 96 | 216
Age, Continuous [Mean (Standard Deviation); unit: years]
  caregiver | 70.6 (11.4) | 69.4 (12.9) | NA (NA) — Data are locked
  care-recipient | 80.4 (6.7) | 80.9 (7.2) | NA (NA) — Data are locked
Gender [Number; unit: participants] — These are care recipients
  participants
    Female | 8 | 6 | 14
    Male | 52 | 42 | 94
Gender [Number; unit: participants] — These are caregivers
  participants
    Female | 49 | 38 | 87
    Male | 11 | 10 | 21
Region of Enrollment [Number; unit: participants]
  United States | 120 | 96 | 216
Physical Self Maintenance Scale [Mean (Standard Deviation); unit: Units on a scale] — Scores range from 6 - 30 with higher scores indicating greater disability
  Units on a scale | 14.6 (4.3) | 15.1 (4.0) | NA (NA) — Data are locked
Mini Mental State Exam [Mean (Standard Deviation); unit: Units on a scale] — Scores range from 0 - 30 with lower scores representing greater cognitive impairment
  Units on a scale | 12.4 (6.6) | 13.0 (6.9) | NA (NA) — Data are locked
Functional Activities Questionnaire [Mean (Standard Deviation); unit: Units on a scale] — Scores range from 0 - 30 with higher scores representing greater disability
  Units on a scale | 25.8 (4.1) | 26.4 (3.1) | NA (NA) — Data are locked

OUTCOME MEASURES:

1. Primary Outcome: Caregiver Strain
Description: Caregiver Strain was measured by the MBRC Caregiver Strain Index; scores ranged from 0 - 15 with higher scores indicating more strain.
Time Frame: 3 months after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Checklist: non-intervention group received conventional home safety checklist
Arm/Group | Home Safety Toolkit | Checklist
Number analyzed (Participants) | 60 | 48
units on a scale | 5.95 (3.17) | 6.96 (3.86)
Statistical Analysis 1: Comparison: Home Safety Toolkit vs Checklist; Test type: Superiority or Other; p < 0.0001, MANCOVA

2. Secondary Outcome: Care Recipient Risky Behaviors and Accidents
Description: The Risky Behavior Checklist listed common risky behaviors and accidents exhibited by care recipients with dementia based on previous research. Potential scores ranged from 0 - undetermined. The maximum score is undetermined because the measure represents the caregiver count of the number of times an incident occurred. In this study, sum scores ranged from 0 - 180.
Time Frame: 3 months after baseline
Measure: Mean (Standard Deviation); unit: number of risky behaviors and accidents
Groups:
- Checklist: Conventional home safety checklist
Arm/Group | Home Safety Toolkit | Checklist
Number analyzed (Participants) | 60 | 48
number of risky behaviors and accidents | 33.95 (32.57) | 37.44 (37.04)
Statistical Analysis 1: Comparison: Home Safety Toolkit vs Checklist; Test type: Superiority or Other; p < .0001, MANCOVA

3. Primary Outcome: Caregiver Self-efficacy
Description: Caregiver self-efficacy was measured by the Revised Checklist for Caregiving Self-Efficacy; the scale consists of 17 items which are rated from 0 - 100% confidence. The total score is summed from these percentages and ranges from 0 - 1700 where higher scores indicate a higher level of confidence.
Time Frame: 3 months after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Home Safety Toolkit | Conventional Safety Checklist
Number analyzed (Participants) | 60 | 48
units on a scale | 1350.30 (197.18) | 1305.65 (203.36)
Statistical Analysis 1: Comparison: Home Safety Toolkit vs Conventional Safety Checklist; Test type: Superiority or Other; p = .002, MANCOVA

ADVERSE EVENTS:
Time Frame: The caregiver reported events to the investigator during 3 months of study participation.
Groups:
- Home Safety Toolkit:Care Recipients: Intervention group receives home safety tool-kit with education and self-efficacy materials to promote competence to make home safety modifications.
  Home Safety Toolkit: Health literacy-verified booklet and home safety items to promote competence to make home safety modifications.
- Checklist:Care Recipients; Checklist:Caregivers: Control group receives conventional list of home safety recommendations
- Home Safety Toolkit:Caregivers: Intervention group receives home safety tool-kit with education and self-efficacy materials to promote competence to make home safety modifications.
Arm/Group | Home Safety Toolkit:Care Recipients | Checklist:Care Recipients | Home Safety Toolkit:Caregivers | Checklist:Caregivers
Serious Adverse Events (participants affected / at risk) | 2/70 | 0/57 | 0/70 | 0/57
Other Adverse Events (participants affected / at risk) | 8/70 | 8/57 | 0/70 | 1/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Home Safety Toolkit:Care Recipients (N=70) | Checklist:Care Recipients (N=57) | Home Safety Toolkit:Caregivers (N=70) | Checklist:Caregivers (N=57)
Death (General disorders) | 2 | 0 | 0 | 0 — Care receivers (frail elderly persons with alzheimer's disease) died in sleep during study but unrelated to study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home Safety Toolkit:Care Recipients (N=70) | Checklist:Care Recipients (N=57) | Home Safety Toolkit:Caregivers (N=70) | Checklist:Caregivers (N=57)
Unanticipated hospitalization (General disorders) | 8 (8) | 8 (8) | 0 (0) | 1 (1) — Care recipient Arms are frail elderly persons with Alzheimer's disease; in Caregiver Arms, spousal caregivers are also frail and prone to hospitalization, requiring withdrawal from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No